CLINICAL TRIAL: NCT01604499
Title: Building on a Point-of-purchase Intervention to Encourage Healthy Food Choices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Anne N. Thorndike, MD, MPH, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011D004784
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Food Labeling
Keywords: Healthy eating; Incentives; Feedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Feedback only (Experimental): Subjects receive feedback letters about the proportion of green, yellow, and red purchases in the cafeteria per month with comparisons to "all employees" and to the "healthiest employees eaters"
  Interventions: Behavioral: Feedback letters
- Feedback plus incentives (Experimental): Subjects receive feedback letters plus small incentives to increase healthy (green-labeled) purchases in the next month
  Interventions: Behavioral: Feedback plus incentives
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Feedback letters — Subjects receive feedback letters about the proportion of green, yellow, and red purchases in the cafeteria per month with comparisons to "all employees" and to the "healthiest employees eaters"
  Arms: Feedback only
Behavioral: Feedback plus incentives — Subjects receive feedback letters plus small incentives to increase healthy (green-labeled) purchases in the next month
  Arms: Feedback plus incentives

SUMMARY:
This study builds on the framework of a previously implemented color-coded food labeling intervention in a hospital cafeteria by testing the incremental effectiveness of providing employees with individual feedback and incentives for increasing healthy purchases in a 3-arm randomized controlled trial. The investigators hypothesize that employees assigned to receive feedback will increase healthy purchases more than employees who receive no contact and that employees who receive feedback plus incentives will increase healthy purchases more than those who receive feedback alone.

ELIGIBILITY:
Inclusion Criteria:

* Employee at Massachusetts General Hospital who uses a cafeteria debit card to pay for cafeteria purchases

Exclusion Criteria:

* Employees who do not have a cafeteria debit card
* Employees with cafeteria debit card but who use it fewer than 3 times a month for the 3 months prior to start of trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2672 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Employee purchases of healthy (green-labeled) items | 6 months

SECONDARY OUTCOMES:
Employee purchases of unhealthy (red-labeled) items | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne N Thorndike, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Thorndike AN, Riis J, Levy DE. Social norms and financial incentives to promote employees' healthy food choices: A randomized controlled trial. Prev Med. 2016 May;86:12-8. doi: 10.1016/j.ypmed.2016.01.017. Epub 2016 Jan 29. PMID 26827617